CLINICAL TRIAL: NCT06657508
Title: Real-World Evaluation of Continuous Glucose Monitoring Data in People With Diabetes and End-Stage Renal Disease Receiving Dialysis
Brief Title: Continuous Glucose Monitoring in People With Diabetes on Dialysis
Acronym: RECORD
Status: Recruiting | Type: Observational
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: 24046
Record Dates: First submitted 2024-10-23; First posted 2024-10-24 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Diabetes Mellitus; End-Stage Renal Disease
Keywords: Diabetes mellitus; End-stage renal disease; End-stage kidney disease; Dialysis; Haemodialysis; Peritoneal dialysis; Kidney replacement therapy; Continuous Glucose Monitoring; Glucose fluctuations
MeSH Terms: conditions — Diabetes Mellitus; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Continuous glucose monitoring is a sensor, which monitors glucose levels continuously throughout the day. In people with diabetes, especially those treated with insulin, this sensor helps guide the amount of treatment (such as insulin) required to maintain glucose within target.

In dialysis, the glucose levels and insulin needs can change a lot because of the kidney failure and dialysis treatments.

The goal of this observational study is to describe the changes in glucose during and in between dialysis sessions over two weeks by using continuous glucose monitoring. The study will also explore whether there is a relationship between the trend of the glucose and fluid level changes during and in between dialysis treatments. Also, the study will assess whether there is a relationship between glucose levels and several long-term outcomes, such as admissions to the hospital, for up to five years.

DETAILED DESCRIPTION:
This is a single-centre observational prospective study, which involves existing users of NHS funded continuous glucose monitoring (CGM) with insulin-treated diabetes mellitus (DM) and end-stage renal disease (ESRD) established on dialysis.

CGM is the standard of care for glucose monitoring in all people with type 1 DM and specific groups with type 2 DM in the United Kingdom.

The study aims to evaluate the association between glucose levels in people with diabetes who are on dialysis with short- and long-term clinical outcomes.

The study will address the following hypotheses:

1. Dialysis causes fluctuation in CGM glucometrics during dialysis and in between dialysis periods.
2. Dysglycaemia is associated with adverse short- and long-term outcomes in people with diabetes who are on dialysis.

The primary objective of the study is to describe glucose levels in the intradialytic and interdialytic periods, by accessing CGM-derived glucometrics over 2 weeks.

The secondary objectives of the study are as follows:

Short term outcomes:

* To understand the impact of dialysis on CGM glucometrics in intradialytic and interdialytic periods (maintenance haemodialysis or peritoneal dialysis) by using raw glucose data combined across multiple different sensors
* To investigate the association of glycaemic control (CGM data and HbA1c) with:

  * Ultrafiltration volume (assessed via body weight change in the intradialytic period)
  * Body composition (assessed by bioelectrical impedance analysis)
  * Blood pressure

Long term outcomes:

* To investigate the association of CGM metrics (intradialytic and interdialytic periods and 14- and 90-day data) and HbA1c with long term outcomes (up to 5 years):

  * Mortality
  * Hospital admissions
  * Cardiovascular events (acute myocardial infarction, stroke, acute or decompensated heart failure)
  * New diabetic foot ulcer or peripheral vascular disease requiring intervention or amputations
* To compare CGM measures with HbA1c as a predictor of long-term outcomes as described above

ELIGIBILITY:
Inclusion criteria:

* Age: ≥18 years (no upper age limit)
* People with insulin-treated diabetes who receive NHS funded continuous glucose monitoring as part of their routine clinical care
* Diabetes duration > 6 months
* People with end-stage renal disease established on dialysis (maintenance haemodialysis or peritoneal dialysis)
* Ability to give informed consent

Exclusion criteria:

* Participation in other competing studies/clinical trials as determined by the study investigator
* Serious illness or events with life expectancy < 3 months or other significant illness which, in the opinion of the study clinician, precludes involvement

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Outpatient secondary care setting. The study population involves people living with diabetes and end-stage renal disease on dialysis (as per eligibility criteria) attending the Renal Unit at the University Hospitals of Derby and Burton NHS Foundation Trust.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-12-31 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Change in continuous glucose monitoring % time in glucose range [3.9-10.0 mmol/l] between intradialytic and interdialytic periods | From baseline to 2 weeks, over 6 consecutive dialysis sessions

SECONDARY OUTCOMES:
Change in continuous glucose monitoring % time in tight glucose range [3.9-7.8 mmol/l] between intradialytic and interdialytic periods | From baseline to 2 weeks, over 6 consecutive dialysis sessions
Change in continuous glucose monitoring % time above glucose range, level 1 [10.1-13.9 mmol/L] between intradialytic and interdialytic periods | From baseline to 2 weeks, over 6 consecutive dialysis sessions
Change in continuous glucose monitoring % time above glucose range, level 2 [>13.9 mmol/l] between intradialytic and interdialytic periods | From baseline to 2 weeks, over 6 consecutive dialysis sessions
Change in continuous glucose monitoring % time below glucose range, level 1 [3.0-3.8 mmol/l] between intradialytic and interdialytic periods | From baseline to 2 weeks, over 6 consecutive dialysis sessions
Change in continuous glucose monitoring % time below glucose range, level 2 [<3.0 mmol/l] between intradialytic and interdialytic periods | From baseline to 2 weeks, over 6 consecutive dialysis sessions
Change in continuous glucose monitoring average glucose between intradialytic and interdialytic periods | From baseline to 2 weeks, over 6 consecutive dialysis sessions
Change in continuous glucose monitoring % coefficient of variation between intradialytic and interdialytic periods | From baseline to 2 weeks, over 6 consecutive dialysis sessions
Change in continuous glucose monitoring Glucose management indicator (GMI) between intradialytic and interdialytic periods | From baseline to 2 weeks, over 6 consecutive dialysis sessions
Relationship between continuous glucose monitoring metrics and baseline Gold score | From baseline to 2 weeks, over 6 consecutive dialysis sessions
  The Gold score assesses hypoglycaemia awareness
Relationship between continuous glucose monitoring metrics and baseline Diabetes Distress Scale [DDS-17] score | From baseline to 2 weeks, over 6 consecutive dialysis sessions
Relationship between continuous glucose monitoring metrics and baseline Problem Areas in Diabetes [PAID] score | From baseline to 2 weeks, over 6 consecutive dialysis sessions
Relationship between continuous glucose monitoring metrics and baseline Glucose Monitoring Satisfaction Survey [GMSS] score | From baseline to 2 weeks, over 6 consecutive dialysis sessions
Relationship between continuous glucose monitoring metrics and baseline Hypoglycaemia Fear Survey-Version II Worry scale [HFS-II W] score | From baseline to 2 weeks, over 6 consecutive dialysis sessions
Relationship between continuous glucose monitoring metrics and baseline Integrated Palliative Outcome Score [IPOS]-renal score | From baseline to 2 weeks, over 6 consecutive dialysis sessions
Relationship between continuous glucose monitoring metrics and baseline Dialysis Thirst Inventory questionnaire score | From baseline to 2 weeks, over 6 consecutive dialysis sessions
Relationship between glucose outcomes and body composition measures on dialysis days assessed by bioelectrical impedance analysis | From baseline to 2 weeks, over 6 consecutive dialysis sessions
  Glucose outcomes include 14- and 90- day continuous glucose monitoring metrics at baseline, intradialytic and interdialytic continuous glucose monitoring metrics, baseline HbA1c
Relationship between glucose outcomes and ultrafiltration volume during dialysis sessions assessed via body weight changes in the intradialytic period | From baseline to 2 weeks, over 6 consecutive dialysis sessions
  Glucose outcomes include 14- and 90- day continuous glucose monitoring metrics at baseline, intradialytic and interdialytic continuous glucose monitoring metrics, baseline HbA1c
Relationship between glucose outcomes and changes in blood pressure in the intradialytic period | From baseline to 2 weeks, over 6 consecutive dialysis sessions
  Glucose outcomes include 14- and 90- day continuous glucose monitoring metrics at baseline, intradialytic and interdialytic continuous glucose monitoring metrics, baseline HbA1c.
  Changes in blood pressure are assessed by measuring blood pressure prior to and post dialysis sessions
Association between glucose outcomes and mortality | From baseline to 5 years
  Glucose outcomes include 14- and 90- day continuous glucose monitoring metrics at baseline, baseline HbA1c, intradialytic and interdialytic continuous glucose monitoring metrics, 14- and 90- day continuous glucose monitoring metrics and HbA1c at month 3, 6, 9 and 12
Association between glucose outcomes and hospital admissions | From baseline to 5 years
  Glucose outcomes include 14- and 90- day continuous glucose monitoring metrics at baseline, baseline HbA1c, intradialytic and interdialytic continuous glucose monitoring metrics, 14- and 90- day continuous glucose monitoring metrics and HbA1c at month 3, 6, 9 and 12
Association between glucose outcomes and cardiovascular outcomes | From baseline to 5 years
  Glucose outcomes include 14- and 90- day continuous glucose monitoring metrics at baseline, baseline HbA1c, intradialytic and interdialytic continuous glucose monitoring metrics, 14- and 90- day continuous glucose monitoring metrics and HbA1c at month 3, 6, 9 and 12.
  Cardiovascular outcomes include acute myocardial infarction, stroke, acute or decompensated heart failure
Association between glucose outcomes and new diabetic foot ulcer requiring intervention or amputation | From baseline to 5 years
  Glucose outcomes include 14- and 90- day continuous glucose monitoring metrics at baseline, baseline HbA1c, intradialytic and interdialytic continuous glucose monitoring metrics, 14- and 90- day continuous glucose monitoring metrics and HbA1c at month 3, 6, 9 and 12
Association between glucose outcomes and new peripheral vascular disease requiring intervention or amputation | From baseline to 5 years
  Glucose outcomes include 14- and 90- day continuous glucose monitoring metrics at baseline, baseline HbA1c, intradialytic and interdialytic continuous glucose monitoring metrics, 14- and 90- day continuous glucose monitoring metrics and HbA1c at month 3, 6, 9 and 12

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals of Derby and Burton, Derby, United Kingdom

IPD SHARING:
Plan to Share IPD: No